CLINICAL TRIAL: NCT03481465
Title: Searching for Early Biomarkers of Long-term Hepatic, Metabolic and Endothelial Dysfunction in Non-affective Psychosis. A 10-year Follow-up Study
Brief Title: Searching for Early Biomarkers of Long-term Hepatic, Metabolic and Endothelial Dysfunction in Non-affective Psychosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Instituto de Investigación Marqués de Valdecilla (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Other Study IDs: HEP_10PAFIP
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia; Psychosis; Metabolic Syndrome
Keywords: Biomarkers; Hepatic dysfunction; Metabolic dysfunction; Endothelial dysfunction; Antipsychotics; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Metabolic Syndrome; Liver Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate, at long-term, the occurrence of liver disease and cardio-vascular risk, in a sample of patients diagnosed with first episode of non-affective psychosis.

DETAILED DESCRIPTION:
Schizophrenia is a severe brain disorder with an excess mortality and reduced life expectancy. It has been proposed that around 60% of this excess mortality is due to physical pathology, mostly cardio-metabolic disorders. In addition to the deleterious effects of hypercaloric diet and sedentary lifestyle, the use of antipsychotic medication has itself a significant effect on metabolism. The metabolic disturbances described related to antipsychotic exposure include weight gain and obesity, dyslipemia, and insulin-resistance or new onset diabetes mellitus, representing cardio-metabolic risk factors leading to cardio-vascular events at the long-run. Some of these metabolic disturbances have been described as relevant factors for non-alcoholic fatty liver disease (NAFLD) development. NAFLD is accepted to be the hepatic component of the metabolic syndrome, and it has been described as an independent cardiovascular risk factor. A recent study by our group found a significant increase in the prevalence of hepatic steatosis after 3 years of antipsychotic treatment in a sample of patients with psychosis. Other studies proposed that there is a link between NAFLD and severe cardio-vascular disease that may be early predicted through peripheral microvascular system signs (endothelial dysfunction). Interestingly, recent studies have shown the presence of endothelial dysfunction in psychosis, probably related to antipsychotic-exposure. In summary, the investigators consider of relevance the study of a possible interrelation between metabolic syndrome, NAFLD, and endothelial dysfunction, at long-term, and their probable correlation with antipsychotic exposure.

Based on the available scientific evidence, the investigators hypothesize that the long-term exposure to antipsychotic medication would be related to liver disease and endothelial dysfunction.

The research project would be implemented as part of a larger prospective longitudinal study on first episode non-affective psychosis, in the First Episode Psychosis Clinical Program (PAFIP). In particular, the project would be part of the "10 PAFIP study", in which those patients that had been included in the PAFIP program 10 years ago will be extensively evaluated (e.g.: clinical, neuroimaging, neuro-psychological, and metabolic evaluations) in order to analyse the long-term progress of the psychosis.

Steatosis and fibrosis indexes would be determined for 10-years time point. For those patients with scores predicting hepatic fibrosis, a full hepatic examination, including elastometry assessment (FibroScan®) with controlled attenuation parameter (CAP) and abdominal ultrasound would be carried out. Moreover, endothelial function would be examined, using EndoPAT2000® and carotid ultrasound evaluation, for those patients turning 10 years since their antipsychotic treatment was firstly prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the First Episode Psychosis Clinical Program (PAFIP) from February 2001 to December 2007.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria of brief psychotic disorder, schizophreniform disorder, schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals included in the Longitudinal Long-term Study of First Episode Psychosis Clinical Program (10-PAFIP) at the University Hospital Marqués de Valdecilla (Santander - Cantabria).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of Non-Alcoholic Fatty Liver Disease (NAFLD) diagnosed by transient elastography (FibroScan®) by spirometry. | 10 years

SECONDARY OUTCOMES:
The presence of endothelial dysfunction measured by EndoPAT2000®. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Javier Vázquez Bourgon, Principal Investigator — Instituto de Investigación Marqués de Valdecilla
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayoral-van Son J, Juncal-Ruiz M, Ortiz-Garcia de la Foz V, Vazquez-Bourgon J, Setien-Suero E, Tordesillas-Gutierrez D, Gomez-Revuelta M, Ayesa-Arriola R, Crespo-Facorro B; PAFIP Research Group. Long-term clinical and functional outcome after antipsychotic discontinuation in early phases of non-affective psychosis: Results from the PAFIP-10 cohort. Schizophr Res. 2021 Jun;232:28-30. doi: 10.1016/j.schres.2021.04.011. Epub 2021 May 16. No abstract available. PMID 34004383
- [Derived] Vazquez-Bourgon J, Ortiz-Garcia de la Foz V, Suarez-Pereira I, Iruzubieta P, Arias-Loste MT, Setien-Suero E, Ayesa-Arriola R, Gomez-Revuelta M, Crespo J, Crespo Facorro B. Cannabis consumption and non-alcoholic fatty liver disease. A three years longitudinal study in first episode non-affective psychosis patients. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Dec 20;95:109677. doi: 10.1016/j.pnpbp.2019.109677. Epub 2019 Jun 20. PMID 31228640